CLINICAL TRIAL: NCT00350480
Title: Treatment of Non-Gestational Acute Uterine BleedingComparing Oral Medroxyprogesterone Acetate and Monophasic Oral Contraceptives Containing Norethindrone and Ethinyl Estradiol
Brief Title: Treatment of Non-Gestational Acute Uterine Bleeding: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uterine Bleeding
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Uterine Hemorrhage; Menorrhagia
Keywords: acute uterine bleeding
MeSH Terms: conditions — Uterine Hemorrhage; Menorrhagia | interventions — Medroxyprogesterone Acetate

INTERVENTIONS:
Drug: Provera
Drug: Combination Birth Control pills

SUMMARY:
To determine the relative efficacy of multidose medroxyprogesterone acetate (MPA, Provera) and a multidose, monophasic combination oral contraceptive in the treatment of hemodynamically stable women with non-gestational, acute uterine bleeding.

DETAILED DESCRIPTION:
Acute uterine bleeding, unrelated to pregnancy, is a relatively common problem that causes many reproductive-aged women to requite emergent medical and/or surgical intervention. Although the traditional approaches have generally been surgical in nature, many practitioners utilize medical methods to arrest the bleeding. However, despite widespread use, there exists a paucity of information regarding the effectiveness, side-effects, and patient satisfaction associated with the commonly-used medical regimens. (b) The purpose of the study is to compare the efficacy of multidose medroxyprogesterone acetate and a multidose, monophasic combined oral contraceptive in the treatment of hemodvnamically-stable women with non-gestational, acute uterine bleeding.

(c) Non-pregnant, hemodynamically-stable, reproductive-aged, women, over the age of IS, who present either to the emergency area or to KP practitioner's offices with acute uterine bleeding, will be considered for eligibility. If, following a full exam and medically appropriate investigations medical management is deemed appropriate, they will be approached by a member of the investigating team for possible inclusion into the study. Following informed consent, patients will be randomized to receive either medroxyprogesterone acetate (20 mg three times daily for 7 days) or monophasic oral contraceptive containing I mg of norethindrone and 35 ug of ethinyl estradiol (three dines daily for seven days). Following the seven days of therapy, those randomized to MPA will continue with 20 mg per day for three weeks while those randomized to oral contraceptives will take one pill per day for three weeks, each completing a total of four weeks of therapy. The primary outcome will be the number of days until cessation of bleeding. Other outcomes measured will include pad and tampon counts, and hemoglobin levels. Chi square tests and student t will be used to evaluate differences between the two treatment groups. The hope is that this study will elucidate on the efficacy of the two regimens.

ELIGIBILITY:
Inclusion Criteria:

Non-pregnant Hemodynamically stable Reproductive-aged women >18 years Present with acute uterine bleeding

Exclusion Criteria:

Pregnant Non-hemodynamically stable <18 years

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2003-04; Study Completion 2005-06

PRIMARY OUTCOMES:
The avoidance of unscheduled surgery in the 28-day follow-up period.
To calculate the time requred from initiation of medical therapy until the cessation bleeding, comparing MPA to monophasic combination oral contraceptive pills.

SECONDARY OUTCOMES:
The assessment of pad and tampon counts.
The assessment of hemoglobin levels, symptoms and side effects (ie: cramping, nausea and bloating) and patient satifaction with medical therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm G Munro, M.D., Principal Investigator — Southern California Permanente Medical Group; Romie Basu, MD, Principal Investigator — Southern California Permanente Medical Group
Locations (1):
- Kaiser Permanente Sunset, Los Angeles, California, United States

REFERENCES:
- [Derived] Munro MG, Mainor N, Basu R, Brisinger M, Barreda L. Oral medroxyprogesterone acetate and combination oral contraceptives for acute uterine bleeding: a randomized controlled trial. Obstet Gynecol. 2006 Oct;108(4):924-9. doi: 10.1097/01.AOG.0000238343.62063.22. PMID 17012455